CLINICAL TRIAL: NCT02600728
Title: Improvement In Gait Performance After Training Based On Declarative Memory Cues In Patients With Parkinson's Disease: A Randomized Clinical Trial
Brief Title: Training Based On Declarative Memory Cues Improved Gait In Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USPNEC006
Record Dates: First submitted 2015-11-04; First posted 2015-11-09 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Gait; cues; memory; training
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental group (EG) (Experimental): The experimental training (ET) consisted of eight gait training sessions, twice a week, using the declarative memory cues strategy (DMCS).
  Interventions: Behavioral: Experimental Training
- control group (CG) (Active Comparator): The control training (CT) consisted of a similar gait training without DMCS.
  Interventions: Behavioral: Control Training

INTERVENTIONS:
Behavioral: Experimental Training — The ET consisted of 3 phases being that the first one (Phase 1) was done only in the first session.
  Phase 1: patients received a short and simple explanation about the deficiency in automatic movement resulting from PD. Following explanation, the patient memorized a sequence of declarative cues. Phase 2: the patient organized a sequence of cues using cards illustrating the subcomponent movements (key movement) involved in taking steps.
  Phase 3: the patient had to train using declarative cues as a gait performance aid through 8 sets follow the instruction "Walk in your ordinary speed. Use the key movements and going to saying each of them while you make them. The declarative cues had to be evoked verbally by the patients themselves, during gait, triggering the corresponding movement.
  Other Names: Declarative memory cues strategy (DMCS)
  Arms: experimental group (EG)
Behavioral: Control Training — The CT consisted of 3 phases, being the first one (Phase 1) was done only in the first session of training, and the other two (Phase 2 and 3) were repeated at each of the 8 sessions.
  Phase 1: Patients received a short and simple explanation about the deficiency in automatic movement resulting from PD.
  Phase 2: Patients received a general verbal attentional instruction of "pay attention to your steps and try to walk as better as you can", before starting the walk.
  Phase 3: motor training of gait, where the patient had to perform 8 sets, following the instruction "Walk in your ordinary speed, paying attention to your steps" in the identical trajectories of ET. Additional instructions or cues were not provided.
  Arms: control group (CG)

SUMMARY:
Deficits in automatic motor control, characteristic of Parkinson's disease (PD), contribute to progressive impairment in gait performance. The use of declarative memory cues in order to promote the engagement of attention and activation of the next movement in gait may minimize the consequences of lack of automatic control. The purpose of this study is to verify the long-term efficiency of a new strategy based on declarative memory cue to improve the gait performance and independence in daily life activities (DLA) in patients with PD.

DETAILED DESCRIPTION:
Background: Deficits in automatic motor control, characteristic of Parkinson's disease (PD), contribute to progressive impairment in gait performance. The use of declarative memory cues in order to promote the engagement of attention and activation of the next movement in gait may minimize the consequences of lack of automatic control.

Objectives: To verify the long-term efficiency of a new strategy based on declarative memory cue to improve the gait performance and independence in daily life activities (DLA) in patients with PD.

Design: Parallel prospective, single blind, randomized clinical trial. Setting: Brazilian Parkinson Association. Participants: Forty-four patients with PD in stages 2-3 of disease evolution according to Hoehn and Yahr Classification Interventions: The experimental training (ET) consisted of eight gait training sessions, twice a week, using the declarative memory cues strategy (DMCS). The control training (CT) consisted of a similar gait training without DMCS.

Primary outcome measure: Gait performance in terms of speed and stride length. Secondary outcome measure: Independence in DLA according to Section II of the Unified Parkinson's Disease Rating Scale.

Randomization: Participants were randomized into a control group (CG), which performed the CT, and an experimental group (EG), which performed the ET, through blinded drawing of names.

Statistical analysis: The gait performance and ADL independence before, 2 and 60 days after the end of training were compared for CG and EG using Repeated-measures analysis of variance (RM-ANOVA).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic Parkinson's disease according to the UK Brain Bank criteria;
* in stage 2-3 of the disease evolution according to the Hoehn and Yahr;
* treated with levodopa or its synergists;
* capable to ambulate independently indoors without aid;
* referring 5 to 15 years of education;
* good visual and auditory acuity.

Exclusion Criteria:

* presence of other neurological (excluding PD), orthopedic or cardiopulmonary problems;
* visual and auditory deficiency;
* dementia [assessed by the Mini Mental State Examination (MMSE), cut-off 23];
* depression [according to the Geriatric Depression Scale (GDS-15), cut-off 6]
* participation in other physical therapy training.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
gait speed | up to 3 months
  The first primary outcome was the gait speed (m/s). Patients were asked to walk in a straight trajectory of 20 meter following the sole instruction "upon the go signal, walk as fast as possible at the line and stop". The speed was calculated based on the time to walk 20 meters timed using a digital chronometer.
stride length on gait | up to 3 months
  The second primary outcome was the stride length (cm) on gait. Patients were asked to walk in a straight trajectory of 20 meter following the sole instruction "upon the go signal, walk as fast as possible at the line and stop". The number of steps was measured using a pedometer.

SECONDARY OUTCOMES:
Independence in activities of daily living (ADL) | up to 3 months
  The secondary outcome was independence in activities of daily living (ADL), assessed by Section II of the Unified Parkinson Disease Rating Scale (UPDRS-II). This section includes 12 questions (items 5 to 16) on patient's performance in ADL. Among these questions, two investigate gait performance (frequent fall due to freezing; inability to walk ), with scores ranging from zero (normal) to 4.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elisa P Piemonte, PhD, Principal Investigator — Department of Physiotherapy, Communication Science & Disorders, Occupational Therapy, School of Medicine, University of São Paulo
Locations (1):
- Department of Physiotherapy, Communication Science & Disorders, Occupational Therapy, School of Medicine, University of São Paulo, São Paulo, São Paulo, Brazil